CLINICAL TRIAL: NCT01445158
Title: Pilot Study of Educational Interventions in Pediatric Hematopoietic Stem Cell Donors to Increase Knowledge of Donation and Transplantation Procedures
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070086; 07-C-0086; NCT00445380 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Normal Donors
Keywords: ShopTalk; Comprehension; Donors; Education; Stem Cell Transplant; Sibling Donor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: bone marrow or stem cell donors ages 10 to 15
- 2: bone marrow or stem cell donors ages 16 to 26

SUMMARY:
Background:

* Hematopoietic Stem Cell Transplant (HSCT) represents the second most frequent major organ transplant in the United States.
* Pediatric 1st degree stem cell donors can experience a variety of psychological difficulties before and after donation with those who feel they are not adequately prepared for possible complications following stem cell donation and transplant describing negative emotions.
* The importance of preparation for children undergoing medical procedures has long been recognized in the field of pediatric psychology

Objectives:

* To assess how prepared pediatric donors are for stem cell donation by assessing their knowledge about stem cell transplants, and to assess their anxiety at different stages of the donation process.
* To assess the effectiveness of a workbook and a board game as tools for conveying information on donation and transplantation to donors.
* To identify donors who may require additional preparation before stem cell collection.
* To explore the relationship between donor knowledge and anxiety symptoms.

Eligibility:

-Stem cell donors ages 10 to 26 years of age

Design:

* Participant s baseline knowledge and anxiety are evaluated.
* Participant s knowledge is reassessed and anxiety evaluated following an information session with the research nurse and doctor about the procedures for stem cell donation and discussion of the consent form for the transplant protocol.
* Participants are separated into two groups. Donors 10 to 15 years of age play a board game; those 16 to 26 years of age are given a workbook on stem cell transplant.
* Participants knowledge and anxiety are reassessed within 24 hours after working with the educational materials and again 1 month later.

DETAILED DESCRIPTION:
Background:

* Hematopoietic Stem Cell Transplant (HSCT) represents the second most frequent major organ transplant in the United States.
* A variety of psychological difficulties in sibling donors post-stem cell donation are reported, including withdrawal, guilt, anger, depression, anxiety, mild to severe psychopathology, and post-traumatic stress symptomatology.
* The importance of preparation for children undergoing medical procedures has long been recognized in the field of pediatric psychology. In previous research, siblings who felt they were not adequately prepared for possible complications following HSCT donation and transplant often described negative emotions.
* Some siblings have reported feeling pressured and coerced to become a donor, while others describe a lack of attention to their physical fears associated with donation and their psychological concerns.
* No prospective studies examining educational tools and transplant knowledge in sibling stem cell donors are currently available.

Objectives:

* To assess pediatric 1st degree stem cell donor comprehension of transplant procedures and compare knowledge prior to educational interventions (pre and post-consent informational session) to knowledge following educational interventions.
* To assess the effectiveness of a workbook intervention as a learning tool for conveying information on stem cell donation and transplantation to pediatric donors.
* To assess the effectiveness of a board game intervention (ShopTalk) as a learning tool for conveying information on stem cell donation and transplantation to pediatric donors.
* To identify donors who may require additional preparation prior to stem cell collection.
* To measure donor anxiety pre and post the educational intervention and stem cell donation and explore the relationship between donor knowledge and anxiety symptoms.

Eligibility:

* Age: 10 to 26 years of age
* Participants or their parents must consent to participation in active bone marrow and peripheral blood stem cell transplant protocols at the NIH.
* For donors less than 18 years of age, their legal guardian must give informed consent, the donor must give written assent.
* For donors greater than or equal to 18 years of age, ability to give informed consent.
* Participants must understand and read English or Spanish.

Design:

* Baseline knowledge will be assessed following consent.
* Knowledge will be reassessed following the information session for the transplant protocol
* Donors will be stratified into 2 groups by age. Donors ages 10 to 15 will be scheduled the following day to play a game called ShopTalk. Donors ages 16 to 26 will be given a workbook on HSCT specifically designed for 1st degree stem cell donors. Knowledge will be reassessed following the administration of these interventions.
* A follow-up assessment will be administered to all participants 1 month after the post intervention test was administered.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: 10 to 26 years of age.
* Participants or their parents must consent to participation in active bone marrow and peripheral blood stem cell transplant protocols at the NIH.
* For donors less than 18 years of age, their legal guardian must give informed consent, the donor must give written assent.
* For donors greater than or equal to 18 years of age, ability to give informed consent.
* Participants must understand and read English or Spanish.

EXCLUSION CRITERIA:

* Presence of psychiatric or psychological symptoms which in the judgment of the Principal or Associate Investigators would compromise the donor's ability to engage in the intervention or is likely to interfere with the study procedures or results.
* Preciously identified cognitive impairment, which in the judgment of the Principal or Associate Investigators would compromise the donor's ability to understand the educational materials or the board game rules and procedures, and is likely to interfere with the study procedures or results.

Ages: 10 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-06-18 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Assess 1st degree relative stem cell donor comprehension of transplant procedures | Prior to relatives transplant
  results of donor quiz and anxiety assessment

SECONDARY OUTCOMES:
Assess efficacy of workbook intervention as a learning tool | Prior to relatives transplant
  results of final quiz after workbook intervention
Assess effectiveness of a board game as a learning tool | Prior to relatives transplant
  results of final quiz after board game
Measure donor anxiety pre-and post educational intervention and pre- and and post educational intervention and pre and post donation | Prior to relatives transplant
  results of anxiety assessment, administered 1 month from initial post intervention test

CONTACTS AND LOCATIONS:
Overall Officials: Lori Wiener, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lipton JM. Peripheral blood as a stem cell source for hematopoietic cell transplantation in children: is the effort in vein? Pediatr Transplant. 2003;7 Suppl 3:65-70. doi: 10.1034/j.1399-3046.7.s3.10.x. PMID 12603696
- [Background] Grupp SA, Frangoul H, Wall D, Pulsipher MA, Levine JE, Schultz KR. Use of G-CSF in matched sibling donor pediatric allogeneic transplantation: a consensus statement from the Children's Oncology Group (COG) Transplant Discipline Committee and Pediatric Blood and Marrow Transplant Consortium (PBMTC) Executive Committee. Pediatr Blood Cancer. 2006 Apr;46(4):414-21. doi: 10.1002/pbc.20800. PMID 16463346
- [Background] Wiley FM, Lindamood MM, Pfefferbaum-Levine B. Donor-patient relationship in pediatric bone marrow transplantation. J Assoc Pediatr Oncol Nurses. 1984 Summer;1(3):8-14. doi: 10.1177/104345428400100304. No abstract available. PMID 6381691
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0086.html